CLINICAL TRIAL: NCT05283278
Title: Effect of Administration of Combined Enteral Lactoferrin and Probiotic On Invasive Fungal Infections In Preterm Neonates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hebatallah A Shaaban, MD, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Pediatrics Dep-ASU
Record Dates: First submitted 2017-10-17; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Fungal Infection
Keywords: Lactoferrin; Probiotic; Preterm
MeSH Terms: conditions — Mycoses; Premature Birth | interventions — Probiotics

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lactoferrin Bovine group (Active Comparator): Group A (20 preterm neonates) which will receive lactoferrin (100mg/day)
  Interventions: Drug: Lactoferrin Bovine
- Lactoferrin Bovine with probiotics group (Active Comparator): Group B (20 preterm neonates) which will receive lactoferrin (100mg/day) in combination with the probiotic
  Interventions: Combination Product: Lactoferrin Bovine and probiotics
- Placebo group (Placebo Comparator): Group C (40 preterm neonates) which is a placebo group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lactoferrin Bovine — Lactoferrin granules (Pravotin®) in a dose of 100 mg /kg/day starting from birth to the 30th day of life for neonates in group A
  Other Names: Pravotin®
  Arms: Lactoferrin Bovine group
Combination Product: Lactoferrin Bovine and probiotics — Lactoferrin granules (Pravotin®) in a dose of 100 mg /kg/day in combination with the probiotic Lactobacillus Delbrueckii and Lactobacillus Fermentum (Lacteol fort®) given in a dose of 5 billions starting from birth to the 30th day of life for neonates in group B
  Other Names: Pravotin® plus Lacteol fort
  Arms: Lactoferrin Bovine with probiotics group
Other: Placebo — Placebo will be given starting from birth to the 30th day of life for neonates in group C.
  Arms: Placebo group

SUMMARY:
The risk for invasive fungal infections is high in very low birth weight (VLBW) infants (< 1500 g) and highest for infants born at the youngest gestational ages who survive past the immediate postnatal period.

Invasive fungal infections (IFIs) represent an increasing cause of severe morbidity and mortality in most neonatal intensive care units.

Lactoferrin (LF) is secreted by epithelial cells into exocrine fluids: seminal fluid, tears, saliva, uterine secretions, and milk. LF is involved in innate immunity mechanisms with several documented anti-infective properties, including antifungal activity.

Probiotics are microorganisms that are believed to provide health benefits when consumed.

It is possible to adopt measures to modify the flora in our bodies and to replace the harmful microbes by useful microbes.

There are certain commercially available strains of probiotic bacteria from the Bifido bacterium and Lactobacillus genera when taken by mouth in daily doses possess treatment efficacy

DETAILED DESCRIPTION:
Bovine LF alone or in combination of probiotics (Lactobacillus Delbrueckii and Lactobacillus Fermentum) can be used in prevention of invasive fungal infection in preterm neonates admitted to the NICU. So, this randomized interventional study aimed at evaluation of the efficacy and safety of enterally administered bovine LF alone or in combination of probiotics (Lactobacillus Delbrueckii and Lactobacillus Fermentum) in comparison to placebo in preterm neonates, through studying blood culture for fungal infection at enrollment, day 7, 14, 21 and 28 using Sabouraud agar for detecting Candida species and Hichrome agar to detect other fungal types ( primary outcome), and to compare length of hospital stay (LOS), use and duration of drug intake as antibiotics and inotropes, use and duration of mechanical ventilation, rate of increase of enteral feeding, time to reach full enteral intake, signs of feeding intolerance, complete blood count (CBC), C reactive protein (CRP), packed red blood cell transfusion (PRBCs) and mortality between the 3 groups as (secondary outcome).

ELIGIBILITY:
Inclusion Criteria:

* 80 preterm
* ≤ 36 weeks gestational age
* >/ = 72 hours of life

Exclusion Criteria:

1. Nothing per os
2. Congenital anomalies.
3. Suspected inborn error of metabolism.
4. Prophylaxis antifungal drugs

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with invasive fungal infection (IFI) | 12 months
  Efficacy of enteral lactoferrin either alone or in combination with the probiotic Lactobacillus Delbrueckii and Lactobacillus Fermentum in the prevention of invasive fungal infections in preterm infants through analyzing the incidence rates of invasive fungal infection (IFI) in all groups using Sabouraud agar for detecting Candida species and Hichrome agar to detect other fungal types.

SECONDARY OUTCOMES:
Number of patients who received packed RBC in each group | 30 days
  The number of patients who received packed RBC in each group from time of enrollment till the 30th day of life
Days on inotropic support in each group | 12 months
  Define how many days required for inotropic support in each group
Days on mechanical ventilation in each group | 12 months
  Define how many days required for mechanical ventilation support in each group
Days of NICU admission in each group | 12 monthes
  Define how many days patients in each group were admitted in the NICU
Number of participants with Necrotizing enterocolitis in each group | 12 months
  Define the rate of NEC occurrence in each group
Mortality in each group | 12 months
  Define the number of mortality in each group

CONTACTS AND LOCATIONS:
Overall Officials: Hebatallah A Shaaban, MD, Study Director — Doctor
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No